CLINICAL TRIAL: NCT05082441
Title: Efficacy of Liposomal Bupivacaine in Benign Soft Tissue Tumor Resection: A Randomized Controlled Trial
Brief Title: Liposomal Bupivacaine in Benign Soft Tissue Tumor Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samaritan Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB20-050
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Benign Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): Exparel group
  Interventions: Drug: Liposomal bupivacaine
- control (Active Comparator): plain bupivacaine
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — Exparel mixed with bupivacaine to be infiltrated in the subcutaneous region of the wound instead of plain bupivacaine
  Other Names: Experimental
  Arms: experimental
Drug: Bupivacaine Hydrochloride — plain bupivacaine subcutaneous injection as standard of care control
  Other Names: Control
  Arms: control

SUMMARY:
Liposomal bupivacaine (Exparel) has been used as an adjunct to pain management in the perioperative setting. However, the efficacy of the drug has not bewen studied in patients with benign soft tissue tumor resections. The goal of the study is to see if Exparel controls pain and improves functional outcomes for patients after these procedures compared to the current standard Bupivacaine HCL.

DETAILED DESCRIPTION:
Liposomal bupivacaine (Exparel) has been used as an adjunct to pain management in the perioperative setting. However, the efficacy of the drug has not bewen studied in patients with benign soft tissue tumor resections. The goal of the study is to see if Exparel controls pain and improves functional outcomes for patients after these procedures compared to the current standard Bupivacaine HCL.

Patients will be randomly assigned Exparel or Bupivacaine HCL intraoperatively during the tumor resection. The amount administered is based on the size of wound after tumor resection. The patients are then provided a pain diary in which they record the amount of pain medications taken, VAS pain scores, and musculoskeletal and tumor society score (MSTS) for the first week postoperatively.

The study will end once 140 patients have been enrolled. Data will be analyzed comparing morphine equivalents, pain scores, and functional scores between the groups.

ELIGIBILITY:
Inclusion Criteria:

* All benign soft tissue tumors greater than one cubic cm
* Adults 18 years and older

Exclusion Criteria:

* Pregnant females
* Women who are breastfeeding
* Less than 18 years old
* Malignant tumors
* Tumors smaller than 1 cubic cm
* Allergy to Exparel
* Patients who are opioid dependent defined as patients on a long acting narcotic or who take more than 30 morphine equivalents per day
* Allergy to amide anesthetics
* bone tumors
* Patients unable to comply with the study standards and follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Use | first 7 days postoperatively
  Amount of morphine equivalents used for postoperative pain control

SECONDARY OUTCOMES:
Pain Score | First 7 days postoperatively
  VAS pain score

OTHER OUTCOMES:
Musculoskeletal Tumor Society Score (MSTS score) | First 7 days postoperatively
  MSTS score postop compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Regional Medical Center, Corvallis, Oregon, United States